CLINICAL TRIAL: NCT01405560
Title: A Phase III Study to Evaluate the Safety, Tolerability, and Efficacy of MK-7009 When Administered Concomitantly With Peginterferon Alfa-2b and Ribavirin in Japanese Patients With Chronic Hepatitis C Infection Who Were Non-responders to Previous Treatment
Brief Title: Vaniprevir Plus PegIntron®/Ribavirin in Japanese Participants With Chronic Hepatitis C Who Are Non-responders to Previous Treatment (MK-7009-045)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7009-045
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — vaniprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaniprevir 24 Week Arm (Experimental): Participants receive 24 weeks of vaniprevir (300 mg twice daily) with concomitant peg-IFN and RBV treatment
  Interventions: Drug: Vaniprevir; Biological: peg-IFN; Drug: ribavirin

INTERVENTIONS:
Drug: Vaniprevir — Capsules containing 150 mg vaniprevir, orally, two in the morning and two in the evening for 24 weeks
  Other Names: MK-7009
Biological: peg-IFN — Open-label peg-IFN alfa-2b at 1.5 μg/kg once per week, administered subcutaneously (SC) for 24 weeks
  Other Names: PegIntron
Drug: ribavirin — Capsules containing 200 mg RBV, orally, 3 to 5 capsules, dosage based on the participant's weight (600 mg/day to 1000 mg/day), for 24 weeks
  Other Names: REBETOL®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of vaniprevir (300 mg twice daily) given in combination with pegylated interferon alfa-2b (peg-IFN) and ribavirin (RBV) in Japanese participants with chronic hepatitis C (CHC) genotype (GT) 1 who have not responded to previous treatment. The primary efficacy objective is to estimate efficacy of vaniprevir, peg-IFN and RBV for 24 weeks as assessed by the percentage of participants achieving undetectable Hepatitis C Virus ribonucleic acid (HCV RNA) 24 weeks after completion of all study therapy (Sustained Viral Response 24 [SVR24]).

ELIGIBILITY:
Inclusion criteria:

* Japanese participant diagnosed with compensated CHC GT 1
* Absence of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease
* Has received and tolerated treatment with IFN-based therapy (IFN α, IFN β, or peg-IFN) with or without use of ribavirin, but failed to respond to the prior treatment (partial responder or null responder)
* No evidence of cirrhosis

Exclusion criteria:

* Co-infection with human immunodeficiency virus (HIV)
* Positive hepatitis B surface antigen or other evidence of active hepatitis B infection
* Any other condition that is contraindicated or for which caution is required for treatment with peg-IFN or RBV
* Any condition or pre-study laboratory abnormality, or history of any illness, that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs, peg-IFN and RBV, to the participant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09-02 (Actual); Primary Completion 2013-03-29 (Actual); Study Completion 2013-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kumada H, Mochida S, Suzuki F, Chayama K, Karino Y, Nakamura K, Fujimoto G, Howe AY, Ludmerer SW, Mobashery N. Vaniprevir plus peginterferon alfa-2b and ribavirin in treatment-experienced Japanese patients with hepatitis C virus genotype 1 (GT1b) infection: Phase 3 studies. J Gastroenterol Hepatol. 2016 Oct;31(10):1674-1683. doi: 10.1111/jgh.13328. PMID 26936417
- [Derived] Ludmerer SW, Hirano T, Black S, Howe AY, Chang W, Takase A, Nakamura K, Tanaka Y, Kumada H, Hayashi N, Nickle D. HCV evolutionary genetics of SVR versus virologic failure assessed from the vaniprevir phase III registration trials. Antiviral Res. 2016 Jun;130:118-29. doi: 10.1016/j.antiviral.2016.03.004. Epub 2016 Mar 3. PMID 26947564
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-045&kw=7009-045&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese patients 20-70 years old (inclusive) with chronic, compensated, genotype 1 Hepatitis C (HCV) infection and HCV ribonucleic acid (RNA) levels ≥5.0 log IU/mL peripheral blood at screening, who had failed to respond to prior interferon treatment, were recruited from 10 sites in Japan.
Pre-assignment Details: 42 participants were randomized to receive 24 weeks of vaniprevir in combination with 24 weeks of peg-IFN α-2b (peg-IFN) and ribavirin (RBV).
Period: Overall Study
Arm/Group | Vaniprevir 24 Week Arm
Started | 42
Completed | 41
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response (SVR)24
Description: SVR24 was defined as having an undetectable HCV RNA level 24 weeks after completion of all study therapy. The percentage of participants achieving SVR24 were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: 24 weeks after 24 weeks of study therapy (up to 48 weeks)
Population: Full Analysis Set (FAS) population; all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 61.9 [45.6 to 76.4]

2. Primary Outcome: Percentage of Participants With One or More Specific Adverse Events (AEs) of Special Interest During the Study
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also an AE. For this study, safety parameters or AEs of special interest that were identified a priori included serious rash, anemia (anemia plus haemoglobin decreased), neutropenia (neutropenia plus neutrophil count decreased), bilirubin increased and gastrointestinal adverse experiences (vomiting, nausea, and diarrhea). The percentage of participants with ≥1 specific AEs were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 48 weeks)
Population: All Participants Treated (APaT) Population; all participants receiving at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants
  With ≥1 specific AEs | 78.6 [63.2 to 89.7]
  anaemia | 40.5 [25.6 to 56.7]
  bilirubin increased | 7.1 [1.5 to 19.5]
  GI AEs | 52.4 [36.4 to 68.0]
  neutropenia | 40.5 [25.6 to 56.7]

3. Secondary Outcome: Percentage of Participants Achieving SVR12
Description: SVR12 was defined as having an undetectable HCV RNA level 12 weeks after completion of all study therapy. The percentage of participants achieving SVR12 were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: 12 weeks after 24 weeks of study therapy (up to 36 weeks)
Population: FAS population; all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 61.9 [45.6 to 76.4]

4. Secondary Outcome: Percentage of Participants Achieving Rapid Virologic Response (RVR)
Description: RVR was defined as having an undetectable HCV RNA level at Week 4. The percentage of participants achieving RVR were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: At Week 4
Population: FAS population; all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 57.1 [41.0 to 72.3]

5. Secondary Outcome: Percentage of Participants Achieving Complete Early Virologic Response (cEVR)
Description: cEVR was defined as having an undetectable HCV RNA level at Week 12. The percentage of participants achieving cEVR were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: At Week 12
Population: FAS population; all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 95.2 [83.8 to 99.4]

6. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV Ribonucleic Acid (RNA) at the End of Treatment (EOT)
Description: Participants were assessed for undetectable HCV RNA levels at the end of all study therapy. The percentage of participants with undetectable HCV RNA levels at EOT were reported along with corresponding 95% Clopper-Pearson exact confidence intervals for each treatment regimen.
Time Frame: At Week 24
Population: FAS population; all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 95.2 [83.8 to 99.4]

7. Secondary Outcome: Mean Change From Baseline in HCV RNA (Log 10)
Description: HCV RNA levels were assessed at baseline (BL) and during treatment weeks 2, 4, 8, 12, and 24 using the Roche TaqMan HCV assay, and transformed to Log 10 values. HCV RNA values below the limit of reliable quantification (LoQ) or the limit of detection (LoD) at any time point were handled as follows (imputations done for computational purposes): values below the LoQ but above the LoD were imputed with the LoQ minus 0.1; values below the LoD were imputed with the value of 0 Log IU/mL. HCV RNA levels below the LoD were considered "undetectable".
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 24
Population: FAS population; all randomized participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Log IU/ml
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
Log IU/ml
  Change From BL at Week 2 (n=42) | -5.5 (0.6)
  Change From BL at Week 4 (n=42) | -6.1 (0.7)
  Change From BL at Week 8 (n=42) | -6.5 (0.7)
  Change From BL at Week 12 (n=41) | -6.5 (1.0)
  Change From BL at Week 24 (n=39) | -6.6 (0.6)

8. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also an AE.
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 48 weeks)
Population: All Participants Treated (APaT) Population; all participants receiving at least one dose of study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Vaniprevir 24 Week Arm
Number analyzed (Participants) | 42
percentage of participants | 2.4

ADVERSE EVENTS:
Time Frame: From Day 1 (post-dose) through completion of Week 24 Follow-up (up to 48 weeks)
Arm/Group | Vaniprevir 24 Week Arm
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 24 Week Arm (N=42)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 24 Week Arm (N=42)
Anaemia (Blood and lymphatic system disorders) | 12 (16)
Neutropenia (Blood and lymphatic system disorders) | 4 (6)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 14 (15)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 7 (8)
Fatigue (General disorders) | 6 (6)
Influenza like illness (General disorders) | 5 (5)
Injection site erythema (General disorders) | 3 (3)
Injection site reaction (General disorders) | 12 (12)
Malaise (General disorders) | 12 (12)
Pyrexia (General disorders) | 25 (31)
Nasopharyngitis (Infections and infestations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 3 (3)
Bilirubin conjugated increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3)
Blood uric acid increased (Investigations) | 3 (4)
Haemoglobin decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 13 (14)
Platelet count decreased (Investigations) | 14 (14)
White blood cell count decreased (Investigations) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 10 (10)
Headache (Nervous system disorders) | 12 (13)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.